CLINICAL TRIAL: NCT00735410
Title: A Phase III, Multicenter, Uncontrolled, Open-label Study to Evaluate Safety and Immunogenicity of Preservative Free, Inactivated Split Influenza Vaccine, Using the Strain Composition 2008/2009 When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Trivalent Split Influenza Vaccine Using the Strain Composition 2008/2009
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V44P12S; 2008-000887-18
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Seasonal Influenza, Vaccine
Keywords: Influenza vaccine; Seasonal; Split
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — 1 dose of Split influenza vaccine

SUMMARY:
Annual trial for registration influenza vaccine with the strain composition for season 2008/2009

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, mentally competent, willing and able to give informed consent prior to study entry
* available for all the visits scheduled in the study and able to comply with all study requirements
* in good health as determined by: medical history physical examination clinical judgment of the investigator

Exclusion Criteria:

* They Have any serious (in the judgment of the investigator) disease, including but not limited to:

Cancer, except for localized skin cancer Advanced congestive heart failure Chronic obstructive pulmonary disease (COPD) Autoimmune disease (including rheumatoid arthritis) Acute or progressive hepatic disease Acute or progressive renal disease Severe neurological or psychiatric disorder Severe Asthma

* They have a history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g., to ovalbumin, chicken protein, chicken feathers, influenza viral protein neomycin or polymyxin).
* Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting for example from:

receipt of immunosuppressive therapy (any parental or oral cortical steroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study; Receipt of immunostimulants, Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study, Suspected or known HIV infection or HIV-related disease.

* Known or suspected history of drug or alcohol abuse.
* They have a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject;
* Women who are pregnant or woman of childbearing potential unwilling to practice acceptable contraception for the duration of the study (21 days).
* Influenza vaccination or laboratory confirmed influenza within the last 6 months and more than one influenza vaccination within the past 12 months
* Within the past 4 weeks they have received:

another vaccine any investigational agent;

* Any acute or chronic infection requiring systemic antibiotic treatment or antiviral therapy within the last 7 days.
* They have experienced fever (i.e., axillary temperature ≥ 38°C) within the last 3 days
* Simultaneous participation in another clinical study.
* Any condition, which, in the opinion of the investigator, might prevent the subject from participation or interfere with the evaluation of the study objectives.
* Severely obese with Body Mass Index (BMI) > 35
* Site personnel involved in evaluation of safety and their immediate relatives are excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of antibody response to each influenza vaccine antigen, as measured by haemagglutination inhibition (HI) test on Day 0 and on Day 21 | 21 days (-1/+7)

SECONDARY OUTCOMES:
Evaluation of safety of the influenza vaccine | 21 days (-1/+7)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Site 1, 2 and 3, Hessen, Germany